CLINICAL TRIAL: NCT00371384
Title: Effect of Massage on Chronic Low Back Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT001927 (NIH); R01AT001927 (NIH)
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Chronic Low Back Pain (Non-specific, Uncomplicated)
Keywords: massage; back pain; effectiveness
MeSH Terms: conditions — Back Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): structural massage
  Interventions: Procedure: massage
- 1 (Experimental): relaxation massage
  Interventions: Procedure: massage

INTERVENTIONS:
Procedure: massage — UP to 10 massages over 10 weeks

SUMMARY:
This study will evaluate the effectiveness of two types of massage therapy for treating chronic low back pain.

DETAILED DESCRIPTION:
Americans are increasingly seeking care from massage therapists for relief of chronic back pain. However, while initial studies suggest that massage is beneficial for back pain, we have no information about which of the many types of massage is most helpful. We will be conducting a study that compares two distinct therapeutic massage protocols with each other and with usual care for treating chronic back pain. This study is designed to determine which of these massage protocols will be most effective in reducing pain and increasing functionality in people with low back pain. 399 Group Health members with non-specific low back pain lasting at least 3 months will be randomized to one of the two massage groups or to a control group that receives no treatment beyond their usual care. Massage therapists will provide each participant with 10 treatments over 10 weeks. The primary outcomes, function and bothersomeness of low back pain, will be assessed before treatment begins and 10, 26 and 52 weeks after randomization by interviewers who do not know which treatment the participant received. The results of this study will clarify the value of two different types of massage for treating one of the most common, challenging, and expensive health problems plaguing developed countries. The findings will help physicians make informed and confident referrals, consumers and insurers make safe and cost-effective choices, and massage schools make responsible curriculum decisions.

ELIGIBILITY:
Inclusion Criteria:

* 20 through 64 years of age
* members of Group Health Cooperative health plan
* low back pain lasting at least 3 months

Exclusion Criteria:

* non-mechanical causes of back pain (e.g., sciatica, systemic/visceral disease, pregnancy, spondylolisthesis, spinal stenosis, cancer, recent vertebral fracture)
* inappropriate candidate for massage (active open skin lesions, conditions exacerbated by increased circulation, recent strokes or heart attacks, compromised immune system, systemic edema, hypersensitivity to touch or loss of sensation, recent surgery, active contagious infection)
* characteristics complicating the interpretation of findings (e.g., involved with litigation or compensation claim, severe or progressive neurological deficit, back surgery within last 3 years, receiving other back treatment)
* unable to speak or read English
* had massage for any reason in prior 12 months

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 399 (Estimated)
Dates: Start 2006-08; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Dysfunction at 10 weeks | 10 weeks
Symptom bothersomeness at 10 weeks | 10 weeks

SECONDARY OUTCOMES:
Dysfunction at 26 and 52 weeks | 26 and 52 weeks
Symptom bothersomeness at 26 and 52 weeks | 26 adn 52 weeks
Anxiety at 10, 26 and 52 weeks | 10 16 and 52 weeks
Depression at 10, 26 and 52 weeks | 10 26 and 52 weeks
Perceived stress at 10, 26 and 52 weeks | 10 26 and 52 weeks
Fear avoidance at 10, 26 and 52 weeks | 10 26 and 52 weeks
Satisfaction with back care at 10 and 26 weeks | 10 and 26 weeks
General health status (SF-36) at 10, 26 and 52 weeks | 10, 26 and 52 weeks
Disability days at 10, 26 and 52 weeks | 10 26 52 weeks
Medication use at 10, 26 and 52 weeks | 10 26 52 weeks
Adverse experiences at 10 weeks | 10 weeks
Perceptions of massage treatments at 10, 26 and 52 weeks | 10 26 52 weeks
Use and cost of health care services for back pain at 10, 26 and 52 weeks | 10 26 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan C Cherkin, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Center for Health Studies, Seattle, Washington, United States

REFERENCES:
- [Derived] Cherkin DC, Sherman KJ, Kahn J, Wellman R, Cook AJ, Johnson E, Erro J, Delaney K, Deyo RA. A comparison of the effects of 2 types of massage and usual care on chronic low back pain: a randomized, controlled trial. Ann Intern Med. 2011 Jul 5;155(1):1-9. doi: 10.7326/0003-4819-155-1-201107050-00002. PMID 21727288
- [Derived] Cherkin DC, Sherman KJ, Kahn J, Erro JH, Deyo RA, Haneuse SJ, Cook AJ. Effectiveness of focused structural massage and relaxation massage for chronic low back pain: protocol for a randomized controlled trial. Trials. 2009 Oct 20;10:96. doi: 10.1186/1745-6215-10-96. PMID 19843340